CLINICAL TRIAL: NCT01048385
Title: The Effect of Concomitant Co Enzyme Q10 Use on Pregnancy Outcome of IVF
Brief Title: The Effect of Co Enzyme Q10 Together With Fertility Drugs on Pregnancy Outcome of in Vitro Fertilization
Acronym: CoQ10-IVF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A new study had shown that polar body biopsies might negatively effect the implantation potential of the embryo.
Sponsor: University of Toronto (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Robert Casper, Prof., University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CoQ10-IVF
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Aneuploidy; Pregnancy; Miscarriage
Keywords: Mitochondrial dysfunction; Mitochondrial nutrients; Aneuploidy; Meiotic Spindle; Coenzyme Q10; Electron transfer chain
MeSH Terms: conditions — Aneuploidy; Abortion, Spontaneous; Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CoQ10 (Experimental): This group will be treated concomitantly with Coenzyme Q10
  Interventions: Dietary Supplement: Coenzyme Q10 concomitant treatment
- Control (Placebo Comparator): Treated with capsules containing the vehicle.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 concomitant treatment — Coenzyme Q10 concomitant treatment to fertility drugs as part of an IVF treatment
  Other Names: Many different brands
  Arms: CoQ10
Dietary Supplement: Placebo — Treated with capsules containing the vehicle (Sesame oil).
  Arms: Control

SUMMARY:
The goal of our research is to increase live birth rates in infertile women and to reduce the incidence of aneuploidy leading to miscarriage and trisomies. We hypothesize that an age related mitochondrial dysfunction reduces the availability of energy in the oocyte and contributes to abnormal segregation of chromosomes during the meiotic division leading to oocyte aneuploidy. Based on preliminary evidence we have obtained in aged mice, we propose that dietary supplementation with Co enzyme Q10 in older women will improve mitochondrial function in the oocytes, leading to a decrease in chromosomal non-disjunction and resulting in embryos with a normal chromosomal complement. Our primary outcome measure will be determination of oocyte chromosome number by multiplex PCR based assay of polar bodies biopsied at the time of IVF. Outcomes of this proposal will enable us to address the mechanisms of ovarian aging and may explain etiology of decreased fertility in older patients. In addition, our work will add to the feasibility of single embryo transfer, thereby avoiding multiple pregnancies and their associated cost to the health care system and to society.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy of CoQ10 administration with respect to its effect on the rate of aneuploidy of oocytes and cumulative live birth rate.

Study Design This is a prospective randomized placebo controlled study. Study participants will undergo up to 3 cycles as part of this protocol. All clinical assessments will be conducted at the participating infertility clinics.

The study will be organized on an outpatient basis at the Toronto Centre for Advanced Reproductive Technology (TCART). The study will involve 54 women aged 35-43 years undergoing IVF treatment. All women will collect 2 mL of saliva in a 5 mL polyethylene tube for baseline measurement of coQ10 activity by arNOX assay (described below).

Study participants will be randomly assigned to either placebo or COQ10 capsules, (AOR - Advanced Orthomolecular Research Inc. 19 St NE Calgary, Alberta, NHPD registration codes 135307). Study participants will take 600 mg of CoQ10 orally once a day with breakfast or identical placebo capsules for 2 months prior to an IVF cycle and up to 3 cycles if pregnancy does not occur. On cycle day 3, subjects will start the ovarian stimulation for in vitro fertilization while continuing the consumption of the supplements. The controlled ovarian stimulation (COH) will consist of the microdose GnRH agonist flare protocol, which is the clinic's standard protocol for older women. COH will be done using recombinant FSH (Puregon; Schering-Plough Inc.,Mississauga, ON, Canada) or human menopausal gonadotropins (Menopur, Ferring Inc, Oakville, ON, Canada) 150 units twice daily S.C. and Buserelin Acetate ( Superfact, Sanofi-Aventis Canada Inc, Laval, Quebec) 0.05 mg subcutaneously B.I.D, and will continue until the day prior to 10,000 units human chorionic gonadotropin (hCG) (Pregnyl, Organon). The dosage will not be changed and must be maintained for the duration of the study. Both drugs will continue daily until follicular development is considered adequate (at least 3 follicles >17 mm, and the E2 level is acceptable for the number of follicles present) at which time the hCG will be injected to trigger final follicular maturation. Oocyte retrieval will be done 36 hours later by vaginal ultrasound guided needle aspiration and with the use of local anesthesia and mild sedation. At the time of retrieval, subjects will collect 2 mL of saliva, in addition, 2 mL of follicular fluid will be collected from the first follicle aspirated from each ovary for determination of coQ10 activity by arNOX assay. AS it is not possible to measure CoQ10 levels in a single cells (e.g. oocytes), FF represents direct cellular environment that can reflect the metabolical profile of this cell. After retrieval, the oocytes will be fertilized with ICSI in order not to contaminate the maternal DNA during polar body biopsy sample with sperm DNA. On the following day, all the oocytes with 2 pronuclei will undergo a biopsy of one or both polar bodies.

Polar body biopsy The oocyte is then inseminated using the intracytoplasmic sperm injection (ICSI) technique and is kept in culture in an incubator. In order to biopsy the polar body, the oocyte is held by the holding pipette with the polar body at the 11-12 o'clock position. An opening is made in the zona pellucida and a polished glass needle is introduced into the perivitelline space and the polar body is carefully removed.

The embryo transfer is performed on the morning of the third day after egg retrieval.

Polar bodies are washed in droplets of isotonic HEPES-buffered saline and then transferred to hypotonic solution, fixed in methanol: acetic acid on a glass slide, and dehydrated in methanol for further genetic analysis. The whole procedure does not adversely affect either fertilization or cleavage rates in biopsied oocytes, as the polar body is not involved in the above processes.Karyotyping:

The polar bodies will be transferred to the UHN microarray center for chromosome number determination. The analysis will be done with a commercial kit from Advalytix ( Olympus Life Science Research, Munich, Germany). This is a multiplex PCR based kit that provides a fast and accurate count of all 23 chromosomes and is tailored to polar body chromosome count. After 2 days a single embryo with a normal karyotype will be transferred to the uterine cavity under ultrasound guidance using a Cook transfer catheter (Cook, Sidney, Australia). The rest of the viable embryos with a normal karyotype will be frozen (Slow freezing). Luteal support will consist of progesterone suppositories 100mg (Kingsway Pharmacy,Toronto, Ontario Canada) vaginally 3 times a day starting on the day of transfer and will continue for 2 weeks until the end of each cycle when serum beta hCG will be drawn and if pregnant, CoQ10/ placebo will be discontinued. If pregnant, luteal support will continue until 10 weeks gestation. If the patient is not pregnant she will have a cycle of endometrial stimulation with micronized estradiol, followed by progesterone once a sufficient endometrial thickness has been measured. Four days afterwards, 1-2 embryos will be thawed and transferred. Luteal support will include estradiol and progesterone which will be maintained up to 10 weeks if pregnant. These cycles of frozen embryo transfer will be continued as long as there are frozen embryos from the same retrieval.

The study endpoints will be:

1. Primary outcome measure will be the number and percentage of euploid eggs per retrieval
2. Secondary outcome measures will include:

   * Ovarian response
   * Embryo quality
   * Cumulative pregnancy rate / retrieval
   * Cumulative live birth rate / retrieval
   * CoQ10 activity in saliva and follicular fluid by arNOX assay

Coenzyme Q10 assay arNOX is a coenzyme Q10-inhibited, aging-related external NADH oxidase (ECTO-NOX) protein of the cell surface that is also present in sera and saliva. It is capable of superoxide generation measured as superoxide dismutase-inhibited reduction of ferricytochrome c (Oxidaised cytochrome C). arNOX activity of saliva of older individuals is inhibited by coenzyme Q10. The activity first appears after age 30 to a near maximum at about age 55.

arNOX activity is assayed from measurements of superoxide production based on the standard method where reduction of ferricytochrome c by superoxide is monitored from the increase in absorbance at 550 nm with reference at 540 nm. As a further check for the specificity of the arNOX activity, superoxide dismutase (SOD) is added near the end of the assay to ascertain that the rate returned to base line. The assay consists of 150 μl (2 mg/ml) oxidized ferricytochrome c solution and 200 μl of saliva added to 2.5 ml assay buffer (8.06 g NaC1, 0.2 g KC1, 0.18 g Na 2HPO4, 0.26 g KH2PO4, 0.13 g CaCl2, 0.1 g MgCl2, 1.35 g glucose dissolved in 1000 ml deionized water, adjusted to pH 7.4, filtered and stored at 4◦C). Rates are determined using a spectrophotometer in the dual wavelength mode with continuous measurements (over 1 min every 1.5 min). After 45 min, 60 μl (containing 60 units) SOD is added and the assay is continued for an additional 45 min.

Salivary arNOX was found to be a convenient and non-invasive method to monitor arNOX levels in clinical coenzyme Q10 intervention trials with the response levels paralleling those seen with serum and cellular arNOX (Morre and Morre 2008).

Study population

A total of 54 female patients desiring pregnancy will be enrolled in this study at TCART- Toronto Center for Advanced Reproductive Technology. Each subject must meet study inclusion and exclusion criteria

Power calculation:

A total of 54 patients will enter this two treatment parallel-design study. The probability is 90 percent that the study will detect a treatment difference at a two sided with p-value ≤ 0.01, if the true difference between the treatments in aneuploidy rate is 25 %. This is based on the assumption that the standard deviation of the response variable is 0.180.

Assignment to treatment and randomization:

Patients will be assigned in chronological order on the day of study enrollment to a computer generated randomization. Each enrolled participant will receive a pre-assigned package containing either placebo or CoQ10 for the duration of the study. The physician will be blinded as to assignment of the patients. Randomization will be done prior to starting the first cycle.

The investigators will keep a separate record relating the names of the subjects to their code numbers, to allow easy checking of data in subject files when required.

Statistical analysis will be done with student t-test to camper between the treatment and placebo group for all the outcome measures. Power analysis was calculated for alpha < 0.01.

Anticipated outcomes and potential pitfalls. The number of patients needed for the study is reasonable and we do not expect it to be an obstacle. If the results in this study will be to the animal study we should be able to show a significant difference in the number of euploid embryos between the test and control groups, as well as with the other outcome parameters. We have been working for several months with the UHN microarray lab to optimize the use of the Advalytics multiplex PCR kit which currently works very well. We do not expect any problems with this component of the object.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-43 years at the time of enrollment
* Diagnosis of primary infertility

Exclusion Criteria:

* Body mass index (BMI) > 38 kg/m2
* Early follicular phase (day 2-4) serum FSH level > 20 mIU/ml.
* Abnormal uterine cavity as evidenced by sonohysterogram or hysterosalpingography
* Any current use of systemic steroid medication or any infertility treatment within 3 months of study enrollment.
* Any contraindication to being pregnant and carrying a pregnancy to term.
* Contraindication for the use of CoQ10, Superfact, Puregon, hCG, Estrace and Progesterone suppositories.
* Any ovarian or abdominal abnormality that may interfere with adequate TVS evaluation.
* Absence of one or two ovaries
* Clinically relevant systemic disease (e.g., Insulin-dependent diabetes, adrenal dysfunction, organic intracranial lesion, polycystic ovarian syndrome, hyperprolactinemia, or hypothalamic tumor) or serious illness (Neoplasia).
* History (within past 12 months) or current abuse of alcohol or drugs.
* Administration of any investigational drugs within three months prior to study enrollment.
* Any medical condition that may interfere with the absorption, distribution, metabolism or excretion of the study drugs, gastrointestinal diseases, mal absorption syndromes and liver dysfunction
* Unexplained gynecological bleeding.
* Ejaculated sperm is not sufficient for ICSI
* Patient not able to communicate adequately with the investigators and to comply with the requirements of the entire study.
* Abnormal COH screening blood done for both partners, including: prolactin, thyroid stimulating hormone, HIV serology, Hepatitis B and C serology, Rubella, group and screen and syphilis serology prior to participation in study.
* Unwillingness to give written informed consent. Previous entry into this study or simultaneous participation in another clinical trial.
* The concurrent use of any of the following drugs:
* Daunorubicin, Doxorubicin, Blood Pressure Medications, Warfarin, Timolol, atorvastatin, cerivastatin, lovastatin, pravastatin, simvastatin gemfibrozil, tricyclic antidepressant medications (including amitriptyline, amoxapine, clomipramine, desipramine, doxepin, imipramine, nortriptyline, protriptyline, and trimipramine) multivitamins or any vitamin supplementation except Folic acid.

Ages: 35 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of euploid eggs per retrieval | 1 year

SECONDARY OUTCOMES:
Ovarian response | 2 years
Embryo quality | 2 years
Cumulative pregnancy rate/retrieval | 2 years
Cumulative live birth rate/retrieval | 2 years
CoQ10 activity in saliva and follicular fluid by arNOX assay | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Casper, Dr., Principal Investigator — University of Toronto
Locations (1):
- The Toronto Center for Advanced Reproductive Technology, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bentov Y, Esfandiari N, Burstein E, Casper RF. The use of mitochondrial nutrients to improve the outcome of infertility treatment in older patients. Fertil Steril. 2010 Jan;93(1):272-5. doi: 10.1016/j.fertnstert.2009.07.988. Epub 2009 Sep 3. PMID 19732879